CLINICAL TRIAL: NCT01678495
Title: Sonothrombolysis Potentiated by Microbubbles as a Novel Treatment of Acute Ischemic Stroke: a Prospective Randomized Pilot Study
Brief Title: Sonothrombolysis Potentiated by Microbubbles for Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIBSP-SPM-2011-63
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Cerebrovascular Stroke
MeSH Terms: conditions — Stroke | interventions — Sulfur Hexafluoride; High-Energy Shock Waves; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sonothrombolysis + microbubbles (Experimental): rtPA+ sonovue. SonoVue sulphur hexafluoride microbubbles 8 microlitres/ml Powder and solvent for dispersion for injection 1 vial containing 25 mg lyophilized powder to be reconstituted with 5 ml sodium chloride 9 mg/ml (0.9%) solution for injection
  1 pre-filled syringe containing sodium chloride 9 mg/ml (0.9%) solution for injection
  1 Mini-Spike Plus 6/8 (CE 0123) transfer system.
  1 ml of the reconstituted dispersion contains 8 microlitres sulphur hexafluoride microbubbles.
  Interventions: Other: Sulfur hexafluoride + ultrasounds; Drug: Recombinant tissue plasminogen activator
- Standard intravenous thrombolysis (Active Comparator): Patients in thecontrol group will use thehelmetbut without U.S continuous U.S wave emission. Serial monitoring of the status ofrecanalizationaccording to theschedule set will be carried out according to theestablished schedule
  Interventions: Drug: Recombinant tissue plasminogen activator

INTERVENTIONS:
Other: Sulfur hexafluoride + ultrasounds
  Arms: Sonothrombolysis + microbubbles
Drug: Recombinant tissue plasminogen activator

SUMMARY:
It has proposed the use of ST without microbubble treatment in randomized association with both intravenous and intra-arterial thrombolysis, but combined treatment (rtPA + U.S.) associated with MB diagnostic not yet been investigated in a randomized study.

The aim of this study is to evaluate efficacy of the combined treatment (r-rtPA+US+MB) vs the standard rtPA treatment in a randomized study in consecutive patients with acute ischemic stroke.

We expect to demonstrate that the combined treatment (rtPA+US+MB) will be statistically superior to standard treatment in terms of recanalization rate.

ELIGIBILITY:
Inclusion Criteria:

* All acute (<4,5 hours) ischemic stroke patients in the MCA territory (as depicted by head computed tomography CT or suspected by clinical data) with a disabling neurological deficit measurable by National Institute of Health Stroke Scale (NIHSS) score, that in the opinion of treating physicians require and meet accepted criteria of treatment with a standard 0.9 mg/kg dose of iv rtPA.
* A documented occlusion of the middle cerebral artery (MCA) documented by TCD and/or angioCT.
* The patient or the legal representative signs the written consent to participate
* Age > or = 18 years
* No significant improvement before treatment.
* The treatment is initiated within 90 minutes of hospital admission (door-to-needle time < or = 90 minutes)
* There is no limitation regarding the NIHSS score. Scores under 5 are usually considered mild strokes, but they can be treated if the investigator believes that the measured deficit is important enough to cause disability. The investigator should weight benefits and risks when the score is under 5 and above 22.

Exclusion Criteria:

* severe stroke as indicated on baseline CT imaging or by a NIHSS score > 25
* evidence of hemorrhage on noncontrast head computed tomography CT),
* any other standard contraindication for intravenous rtPA therapy,
* primary treatment with intra-arterial thrombolysis,
* Previous Rankin scale score > 1 and NIHSS < 14 or previous Rankin scale score > 2 and NIHSS > or = 14
* Rapidly improving neurological symptoms such that the rate of improvement is expected to result in a NIHSS score of < 4 at randomization
* Coexisting neurological diseases such as dementia or life-threatening illness.
* Seizure at symptom onset
* History or clinical presentation of intracranial hemorrhage, subarachnoid hemorrhage (even with a normal CT), arteriovenous malformation, aneurysm, spinal cord disease or cerebral neoplasm. Incidental meningioma and microbleeds per se are not exclusion criteria.
* Baseline blood glucose concentration less than 50 mg/dL or greater than 400 mg/dl, that cannot be corrected
* Uncontrolled hypertension, defined as systolic blood pressure > 185 mm Hg or diastolic blood pressure > 110 mm Hg on at least two separate occasions at least 10 min apart, or blood pressure that requires aggressive treatment to reduce it to within these limits
* Hereditary or acquired hemorrhagic diathesis
* Another stroke, a serious head injury or major surgery within the previous 3 month
* Platelet count < 100.000/mm3
* Hemorrhagic retinopathy
* Within 10 days of traumatic external heart massage, obstetrical delivery, recent puncture of a non-compressible blood-vessel
* Bacterial endocarditis, pericarditis
* Acute pancreatitis; documented ulcerative gastrointestinal disease during the last 3 months, esophageal varices
* Arterial aneurysm, arterial/venous malformations
* Neoplasm with increased bleeding risk
* Severe liver disease, including hepatic failure, cirrhosis, portal hypertension and active hepatitis
* Major surgery or significant trauma in past 3 months
* Contraindication to CT perfusion: Iodinated contrast allergy, renal insufficiency (elevated serum creatinine above normal laboratory levels at each center), non-collaborative patients, pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-08; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Recanalization rate | 6 h, 24h, and day 90 post treatmente
  The short term efficacy of treatment will be evaluated by recanalization rate at 6 hours control TCD (TIBI score) and at 24 hours by the NIHSS (a > 4 points improvement). As explained, the Rankin scale score will be used to test the efficacy of the treatment at day 90 after stroke onset.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain